CLINICAL TRIAL: NCT00025415
Title: A Phase I Pharmacokinetic Study of STI571 in Patients With Advanced Malignancies and Varying Levels of Liver Dysfunction
Brief Title: Imatinib Mesylate in Treating Patients With Advanced Cancer and Liver Dysfunction
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02418; 01-028; U01CA099168 (NIH); U01CA062505 (NIH); U01CA062491 (NIH); U01CA062502 (NIH); U01CA062487 (NIH); CDR0000068959 (Registry Identifier: PDQ (Physician Data Query)); NCT00025948 (obsolete NCT alias)
Record Dates: First submitted 2001-10-11; First posted 2003-01-27 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2013-02

CONDITIONS: Accelerated Phase Chronic Myelogenous Leukemia; Acute Undifferentiated Leukemia; AIDS-related Peripheral/Systemic Lymphoma; AIDS-related Primary CNS Lymphoma; Anaplastic Large Cell Lymphoma; Angioimmunoblastic T-cell Lymphoma; Atypical Chronic Myeloid Leukemia, BCR-ABL1 Negative; Blastic Phase Chronic Myelogenous Leukemia; Childhood Myelodysplastic Syndromes; Chronic Eosinophilic Leukemia; Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Chronic Myelomonocytic Leukemia; Chronic Neutrophilic Leukemia; Chronic Phase Chronic Myelogenous Leukemia; de Novo Myelodysplastic Syndromes; Essential Thrombocythemia; Extramedullary Plasmacytoma; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Gastrointestinal Stromal Tumor; Intraocular Lymphoma; Isolated Plasmacytoma of Bone; Meningeal Chronic Myelogenous Leukemia; Monoclonal Gammopathy of Undetermined Significance; Myelodysplastic/Myeloproliferative Neoplasm, Unclassifiable; Nodal Marginal Zone B-cell Lymphoma; Polycythemia Vera; Previously Treated Myelodysplastic Syndromes; Primary Central Nervous System Non-Hodgkin Lymphoma; Primary Myelofibrosis; Primary Systemic Amyloidosis; Progressive Hairy Cell Leukemia, Initial Treatment; Prolymphocytic Leukemia; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Acute Myeloid Leukemia; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Hodgkin Lymphoma; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Adult T-cell Leukemia/Lymphoma; Recurrent Cutaneous T-cell Non-Hodgkin Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Mycosis Fungoides/Sezary Syndrome; Recurrent Small Lymphocytic Lymphoma; Refractory Chronic Lymphocytic Leukemia; Refractory Hairy Cell Leukemia; Refractory Multiple Myeloma; Relapsing Chronic Myelogenous Leukemia; Secondary Acute Myeloid Leukemia; Secondary Myelodysplastic Syndromes; Small Intestine Lymphoma; Splenic Marginal Zone Lymphoma; Stage IV Adult Burkitt Lymphoma; Stage IV Adult Diffuse Large Cell Lymphoma; Stage IV Adult Diffuse Mixed Cell Lymphoma; Stage IV Adult Diffuse Small Cleaved Cell Lymphoma; Stage IV Adult Hodgkin Lymphoma; Stage IV Adult Immunoblastic Large Cell Lymphoma; Stage IV Adult Lymphoblastic Lymphoma; Stage IV Adult T-cell Leukemia/Lymphoma; Stage IV Chronic Lymphocytic Leukemia; Stage IV Cutaneous T-cell Non-Hodgkin Lymphoma; Stage IV Grade 1 Follicular Lymphoma; Stage IV Grade 2 Follicular Lymphoma; Stage IV Grade 3 Follicular Lymphoma; Stage IV Mantle Cell Lymphoma; Stage IV Marginal Zone Lymphoma; Stage IV Mycosis Fungoides/Sezary Syndrome; Stage IV Small Lymphocytic Lymphoma; T-cell Large Granular Lymphocyte Leukemia; Unspecified Adult Solid Tumor, Protocol Specific; Untreated Adult Acute Lymphoblastic Leukemia; Untreated Adult Acute Myeloid Leukemia; Untreated Hairy Cell Leukemia; Waldenström Macroglobulinemia
MeSH Terms: conditions — Leukemia, Myeloid, Accelerated Phase; Leukemia, Biphenotypic, Acute; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Blast Crisis; Pdgfra-Associated Chronic Eosinophilic Leukemia; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myelomonocytic, Chronic; Leukemia, Neutrophilic, Chronic; Leukemia, Myeloid, Chronic-Phase; Thrombocythemia, Essential; Gastrointestinal Stromal Tumors; Intraocular Lymphoma; Monoclonal Gammopathy of Undetermined Significance; Myeloproliferative Disorders; Lymphoma, B-Cell, Marginal Zone; Polycythemia Vera; Primary Myelofibrosis; Immunoglobulin Light-chain Amyloidosis; Leukemia, Prolymphocytic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Hairy Cell; Multiple Myeloma; Leukemia, Large Granular Lymphocytic; Waldenstrom Macroglobulinemia | interventions — Imatinib Mesylate

ARMS (1):
- Treatment (imatinib mesylate) (Experimental): Patients receive oral imatinib mesylate daily. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients within each stratum (except normal stratum) receive escalating doses of imatinib mesylate until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity
  Interventions: Drug: imatinib mesylate; Other: pharmacological study

INTERVENTIONS:
Drug: imatinib mesylate — Given orally
  Other Names: CGP 57148; Gleevec; Glivec
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Phase I trial to study the effectiveness of imatinib mesylate in treating patients who have advanced cancer and liver dysfunction

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose and dose-limiting toxicity of imatinib mesylate in patients with advanced malignancies and varying degrees of liver dysfunction.

II. Determine the effects of hepatic dysfunction on the pharmacodynamics and pharmacokinetics of this drug in these patients.

III. Determine the non-dose-limiting toxic effects of this drug in these patients.

IV. Determine the response rate of these patients treated with this drug. V. Correlate the Childs-Pugh classification of hepatic dysfunction with observed toxic effects, pharmacodynamics, and pharmacokinetics of this drug in these patients.

OUTLINE: This is a dose-escalation, multicenter study. Patients are stratified according to liver dysfunction (normal vs mild vs moderate vs severe).

Patients receive oral imatinib mesylate daily. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients within each stratum (except normal stratum) receive escalating doses of imatinib mesylate until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

PROJECTED ACCRUAL: A total of 60 patients will be accrued for this study within 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed surgically incurable solid tumor orhematologic malignancy for which no standard or palliative therapy exists oris no longer effective

  * All tumor types are eligible, including:

    * Chronic myelogenous leukemia or other Philadelphia chromosome-positive leukemia OR
    * Gastrointestinal stromal tumors
* Patients with gliomas that require corticosteroids or anticonvulsants must beon a stable dose and seizure-free for 1 month
* No unstable or untreated (non-irradiated) brain metastases
* Performance status - ECOG 0-2
* Performance status - Karnofsky 60-100%
* More than 3 months
* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* No active hemolysis
* See Surgery
* No evidence of biliary sepsis
* Creatinine normal
* Creatinine clearance at least 60 mL/min
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* Able to swallow pills
* No other uncontrolled concurrent illness that would preclude study participation
* No ongoing or active infection
* No uncontrolled diarrhea
* No psychiatric illness or social situation that would preclude study compliance
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception during and for 6 months after study completion
* At least 24 hours since prior colony-stimulating factors
* No concurrent colony-stimulating factors
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered
* See Disease Characteristics
* See Disease Characteristics
* At least 4 weeks since prior radiotherapy and recovered
* See Disease Characteristics
* At least 10 days since prior placement of shunt for treatment of biliary obstruction
* At least 14 days since prior major surgery
* No prior solid organ transplantation
* No other concurrent investigational agents
* No concurrent therapeutic doses of warfarin for anticoagulation
* No other concurrent investigational or commercial agents or therapies for treatment of this disease
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No concurrent acetaminophen of more than 4,000 mg/day

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2001-08; Primary Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
MTD defined based on the toxicities observed during the first cycle of treatment | 4 weeks
Toxicity evaluation graded according to the NCI common toxicity criteria and relationship to the study drug | Up to 4 years
  Results will be tabulated by liver dysfunction group.

SECONDARY OUTCOMES:
Pharmacokinetic data | Day 1, 2, 3, 4, 15, 16
  Will be analyzed with ADAPT II, and results will be summarized separately for the four study groups. Additionally, results for pharmacokinetic parameters will be related to the measured level of liver dysfunction in exploratory analyses.
Responses | Up to 4 years
  Will be tabulated by liver dysfunction group, and by dose if appropriate.
Child-Pugh Classification | Baseline
  Will be correlated to the toxicities, pharmacokinetic and pharmacodynamic data seen with STI571.

CONTACTS AND LOCATIONS:
Overall Officials: Ramesh Ramanathan, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States